CLINICAL TRIAL: NCT06244901
Title: Community Testing of Wearable Assistance
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Northern Arizona University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 2137424
Record Dates: First submitted 2023-07-13; First posted 2024-02-06 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-01

CONDITIONS: Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Exoskeleton Walking (Experimental): Walking with ankle exoskeleton assistance
  Interventions: Device: Ankle Exoskeleton
- Normal walking (Placebo Comparator): Walking under normal conditions (no exoskeleton)
  Interventions: Other: Normal walking

INTERVENTIONS:
Device: Ankle Exoskeleton — Walking for twenty minutes with a wearable powered robotic ankle exoskeleton on real-world terrain every day for a week.
  Arms: Exoskeleton Walking
Other: Normal walking — Normal walking for twenty minutes on real-world terrain every day for a week.
  Arms: Normal walking

SUMMARY:
This feasibility study looks to evaluate ankle exoskeleton assistance in community settings for individuals with cerebral palsy.

DETAILED DESCRIPTION:
Participants will undergo consent (if not done over the phone), history/physical/activity questionnaire, and orthotic device fitting. Following device fitting, the participants will practice walking with powered assistance.

Next, participants will complete "pre" walking tests with and without the device (order randomized) on a 15-minute pre planned community walk in close proximity with their own home. Distance, time, heart-rate, and perceived exertion will be recorded. The expected duration is 1-2 hours.

Next, participants will be asked to complete (under parental supervision for minors) the pre-determined walking route every day for 1 week with or without ankle exoskeleton assistance (block randomized). Following the first week of independent walking practice, participants will complete "post" walking tests with and without the device on the same walking route. Distance, time, heart-rate, and perceived exertion will be recorded. The expected duration is 1-2 hours.

Participants will then have a 2-6 week washout period.

Following this washout, the pre- and post-assessments will be completed before and after, respectively, another week of identical community walking practice completed under the remaining condition (either exoskeleton or no exoskeleton).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of cerebral palsy
* Gross Motor Function Classification Level I, II, or III
* Able to walk for at least 20 minutes with or without a walking aid
* Able to safely fit into a device configuration and tolerate assistance without knee hyperextension while walking
* Able to provide verbal assent, if appropriate. If the participant is non-verbal, parental interpretation of gesticulation for assent will be used.

Exclusion Criteria:

* Any neurological, musculoskeletal or cardiorespiratory injury, health condition ( including pregnancy), or diagnosis other than cerebral palsy that would affect the ability to walk as directed for short periods of time.
* Participant or parent report that the perspective participant's physician has recommended that they not engage in moderate intensity walking exercise.

Ages: 12 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-10-25 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Walking speed | through study completion, an average of one week
  Change in walking speed (measured in meters per second)

SECONDARY OUTCOMES:
Step length | Through study completion, an average of one week
  Change in step length (measured in meters)
Heart-rate | Through study completion, an average of one week
  Change in heart rate (measured in beats per minute)
Perceived exertion | Through study completion, an average of one week
  Change in perceived exertion (measured on a 1-10 scale)

CONTACTS AND LOCATIONS:
Locations (1):
- Northern Arizona University, Flagstaff, Arizona, United States

IPD SHARING:
Plan to Share IPD: No